CLINICAL TRIAL: NCT00000763
Title: A Phase I Study of TNP-470 in the Treatment of AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 215; 11192 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antineoplastic Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — O-(Chloroacetylcarbamoyl)fumagillol

INTERVENTIONS:
Drug: TNP-470

SUMMARY:
To assess toxicity and determine the MTD of intravenous TNP-470 administered weekly in patients with AIDS-related Kaposi's sarcoma. To assess pharmacokinetics and tumor response of the drug.

Since evidence shows that neovascularization is important in the development of Kaposi's sarcoma, drugs that inhibit angiogenesis, such as TNP-470, may be of benefit in patients with the disease.

DETAILED DESCRIPTION:
Since evidence shows that neovascularization is important in the development of Kaposi's sarcoma, drugs that inhibit angiogenesis, such as TNP-470, may be of benefit in patients with the disease.

Patients are entered at 7 escalating dose levels of TNP-470. (PER AMENDMENT 9/3/96: dose maximum level changed.) Four patients treated at a given dose level must receive at least 4 weeks of therapy before escalation in subsequent cohorts proceeds. If 50 percent of patients at a given dose level experience dose-limiting toxicity, the previous dose is defined as the MTD and an additional two patients are treated at the MTD. Patients receive treatment for 12 weeks, followed by 2 weeks of rest, followed by an additional 12 weeks of treatment. Patients are followed for 12 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT, ddI, ddC, or d4T provided patients have received at least 2 weeks of this therapy prior to study entry. (Combination ddI/ddC is not permitted.)
* MAI prophylaxis.

Required in patients with CD4 count < 200 cells/mm3:

Aerosolized pentamidine, trimethoprim/sulfamethoxazole, or dapsone as PCP prophylaxis.

Patients must have:

* HIV infection.
* Cutaneous Kaposi's sarcoma.
* Life expectancy of at least 3 months.
* Consent of parent or guardian if under 18 years of age.

NOTE:

* This protocol is considered suitable for prison populations.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Peripheral neuropathy (grade 2 or worse).
* Underlying severe or life-threatening infection with bacterial, viral, fungal, or protozoal pathogens.
* Known hypersensitivity to TNP-470, fumagillin, or known related compounds.

PER AMENDMENT 9/3/96:

* Cataracts.

Concurrent Medication:

Excluded:

* Combination therapy with ddI/ddC (although these drugs may be administered alone or in combination with AZT).
* Anticonvulsive medication.
* Steroids.
* Antineoplastic drugs.
* Interferons.
* Systemic or topical anti-Kaposi's sarcoma agents or regimens.
* Suramin.
* Aspirin.
* Warfarin.
* Heparin (including heparin flushes).
* Nonsteroidal anti-inflammatory drugs.
* Investigational status drugs.

Patients with the following prior conditions are excluded:

* History of substantial non-iatrogenic bleeding disorders.
* History of tumor or malignancies other than Kaposi's sarcoma, with the exception of completely resected basal cell skin carcinoma or in situ cervical carcinoma.
* History of seizures within the past 10 years.

PER AMENDMENT 9/3/96:

* History of cataracts.

Prior Medication:

Excluded within 4 weeks prior to study entry:

* Steroids.
* Antineoplastic drugs.
* Interferons.
* Systemic or topical anti-Kaposi's sarcoma agents or regimens.

Excluded within 6 months prior to study entry:

* Suramin.

Unwilling to refrain from unprotected sexual contact or other activities that may result in HIV re-infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Study Completion 1997-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gill PS, Study Chair; Dezube B, Study Chair
Locations (6):
- United States (6):
  - USC CRS, Los Angeles, California
  - Northwestern University CRS, Chicago, Illinois
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York

REFERENCES:
- [Background] Dezube BJ, Von Roenn JH, Holden-Wiltse J, Cheung TW, Remick SC, Cooley TP, Moore J, Sommadossi JP, Shriver SL, Suckow CW, Gill PS. Fumagillin analog in the treatment of Kaposi's sarcoma: a phase I AIDS Clinical Trial Group study. AIDS Clinical Trial Group No. 215 Team. J Clin Oncol. 1998 Apr;16(4):1444-9. doi: 10.1200/JCO.1998.16.4.1444. PMID 9552050
- [Background] Frenkel LM, Wagner LE 2nd, Atwood SM, Cummins TJ, Dewhurst S. Specific, sensitive, and rapid assay for human immunodeficiency virus type 1 pol mutations associated with resistance to zidovudine and didanosine. J Clin Microbiol. 1995 Feb;33(2):342-7. doi: 10.1128/jcm.33.2.342-347.1995. PMID 7714190
- [Background] Pluda JM, Wyvill K, Lietzau J, Figg D, Saville MW, Nguyen BY, Foli A, Bailey J, Cooper M. A phase I trial of TNP-470 (AGM-1470) administered to patients with HIV-associated kaposi's sarcoma (KS). Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:61